CLINICAL TRIAL: NCT00002510
Title: HIGH-DOSE CHEMORADIOTHERAPY FOLLOWED BY RESCUE WITH MOBILIZED AUTOLOGOUS PERIPHERAL BLOOD STEM CELLS IN PATIENTS WITH LOW-GRADE, TRANSFORMED, OR FOLLICULAR LARGE CELL NON-HODGKIN'S LYMPHOMA
Brief Title: Chemotherapy and Radiation Therapy Followed by Peripheral Stem Cell Transplantation in Treating Patients With Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: Fox Chase Cancer Center (Other)
Responsible Party: Temple University Bone Marrow Transplant Program, Temple University Health Systems
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000078066; TUHSC-2049; NCI-V92-0206
Record Dates: First submitted 1999-11-01; First posted 2004-08-23 (Estimated); Last update posted 2010-10-01 (Estimated); Status verified 2010-09

CONDITIONS: Lymphoma
Keywords: Waldenstrom macroglobulinemia; recurrent small lymphocytic lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma
MeSH Terms: conditions — Lymphoma; Waldenstrom Macroglobulinemia; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Follicular | interventions — Filgrastim; Cyclophosphamide; Etoposide; Mesna; Peripheral Blood Stem Cell Transplantation; Radiotherapy

INTERVENTIONS:
Biological: filgrastim
Drug: cyclophosphamide
Drug: etoposide
Drug: mesna
Procedure: peripheral blood stem cell transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage cancer cells. Peripheral stem cell transplantation may allow doctors to give higher doses of chemotherapy and radiation therapy and kill more cancer cells.

PURPOSE: Phase I/II trial to study the effectiveness of etoposide plus radiation therapy followed by peripheral stem cell transplantation in treating patients who have non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the overall and progression-free survival of patients with selected poor-prognosis non-Hodgkin's lymphomas treated with high-dose etoposide and total-body irradiation followed by rescue with peripheral blood stem cells. II. Determine the toxicity of this regimen. III. Evaluate the short-term and long-term engraftment characteristics of patients treated on this regimen.

OUTLINE: Patients who respond on Regimen A and who have no bulk disease greater than 5 cm are treated on Regimen B. Regimen A: Single-Agent Chemotherapy/Stem Cell Mobilization with Urothelial Protection and Growth Factor Therapy. Cyclophosphamide, CTX, NSC-26271; with Mesna, NSC-113891; and Granulocyte Colony Stimulating Factor (Amgen), G-CSF, NSC-614629. Regimen B: Sequential Radiotherapy, Single-Agent Chemotherapy, and Stem Cell Rescue. Total-body irradiation, TBI (equipment not specified); Etoposide, VP-16, NSC-141540; and Peripheral Blood Stem Cells, PBSC.

PROJECTED ACCRUAL: 20 patients will be studied.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Pathologically confirmed non-Hodgkin's lymphomas of the following histologic subtypes: Small lymphocytic Follicular small cleaved cell Follicular mixed cell Follicular large cell (relapsed) Disease in first, second, or third partial remission (25% shrinkage in cross-sectional area of measurable disease) or first, second, or subsequent relapse required Transformed non-Hodgkin's lymphoma eligible, i.e., low-grade lymphoma subsequently transformed to intermediate- or high-grade lymphoma No lymphosarcoma cell leukemia

PATIENT CHARACTERISTICS: Age: 16 to 65 Performance status: Karnofsky 80-100% Hematopoietic: WBC at least 5,000/mm3 (polys at least 2,000/mm3) Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 2.0 mg/dL SGOT no greater than 2 times normal Renal: Creatinine no greater than 1.8 mg/dL Cardiovascular: LVEF at least 50% Pulmonary: FVC greater than 1.5 liters FEV1 greater than 1.2 liters MVV greater than 50 liters DLCO greater than 12 mL/min pO2 greater than 70 mm Hg on room air Other: No other serious psychiatric, neurologic, or medical illness

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: Not specified Endocrine therapy: Not specified Radiotherapy: Less than 3,500 cGy prior irradiation to the mediastinum, lungs, or spinal cord Surgery: Not specified

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1992-04; Primary Completion 2001-06 (Actual); Study Completion 2001-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas R. Klumpp, MD, Study Chair — Fox Chase Cancer Center
Locations (1):
- Temple University Cancer Center, Philadelphia, Pennsylvania, United States